CLINICAL TRIAL: NCT07180446
Title: Predicting Exercise-Induced Insulin Sensitivity With AI: Butyrate Supplementation as a Therapy for Exercise-Resistant Individuals
Brief Title: Can Gut Bacteria Predict Who Benefits Most From Exercise? A Gut Supplement to Help Exercise Non-Responders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Elisa Marroquin, Assistant Professor, Texas Christian University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Exercise - Gut Microbiome
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Obesity &Amp; Overweight
Keywords: Butyrate; Gut Microbiome; Exercise; Cardiovascular; Insulin; Gut Microbiota
MeSH Terms: conditions — Obesity; Overweight; Motor Activity; Insulin Resistance | interventions — Butyrates

STUDY DESIGN:
Intervention Model Description: Interventional Study Model:
  Type: Interventional (Clinical Trial)
  Design: Single-group assignment (one-arm study)
  Model: Pretest-Posttest Design
  Allocation: Non-randomized
  Masking: None (Open Label)
  Primary Purpose: Treatment / Mechanistic
  Time Perspective: Prospective
  Study Duration: 12 weeks
  Intervention Type:
  Behavioral: Supervised cardiovascular exercise (progressively increasing intensity over 12 weeks)
  Dietary Supplement: Sodium butyrate (oral capsules, 6 per day, taken during weeks 8-12)
  Description:
  Participants will undergo a 12-week exercise intervention. During the final 4 weeks, they will additionally receive sodium butyrate supplementation. The model uses repeated measures to assess changes in insulin sensitivity, gut microbiome composition, and body composition before and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Participants will undergo a 12-week exercise intervention. During the final 4 weeks, they will additionally receive sodium butyrate supplementation. The model uses repeated measures to assess changes in insulin sensitivity, gut microbiome composition, and body composition before and after the intervention.
  Interventions: Behavioral: Cardiovascular Exercise; Dietary Supplement: Butyrate

INTERVENTIONS:
Behavioral: Cardiovascular Exercise — Participants will complete a 12-week supervised cardiovascular exercise program at the TCU Recreation Center. Exercise will occur 5 days per week, beginning with 30 minutes per session and progressing to 60 minutes. Intensity will start at 50% of estimated maximal heart rate and gradually increase to 80% by week 8, remaining at that level through week 12. Exercise modalities may include treadmill walking/running, rowing, elliptical, or cycling, based on participant preference and fitness level. Certified trainers will supervise all sessions to ensure safety, proper technique, and adherence to the intensity targets. Participants will wear ActiGraph heart rate monitors to verify exercise intensity throughout the intervention.
Dietary Supplement: Butyrate — Participants will take a dietary supplement containing sodium butyrate during the final 4 weeks (weeks 8-12) of the 12-week intervention. The supplement will be provided in capsule form, with participants instructed to take six capsules per day-two with each meal. This daily dose is equivalent to 3.6 g of butyric acid, which provides 939 mg of sodium, delivered as sodium butyrate. The supplement is intended to support gut health and potentially enhance insulin sensitivity in individuals who do not respond to exercise alone. Participants will receive a 4-week supply during their 8-week study visit, along with instructions for proper use and monitoring of any side effects.

SUMMARY:
The goal of this clinical trial is to learn how gut bacteria affect the way the body responds to exercise, especially how the body uses insulin. It also aims to learn if a supplement called sodium butyrate can help people who don't respond well to exercise alone.

The main questions it aims to answer are:

* Does exercise improve how the body uses insulin in male participants who have overweight or obesity?
* Can gut bacteria predict who will benefit most from exercise?
* Does sodium butyrate help improve insulin response in people who don't respond to exercise alone?

Participants will:

* Exercise 5 days a week for 12 weeks under supervision
* Take sodium butyrate (a natural gut health supplement) daily for the last 4 weeks of the program
* Provide blood and stool samples at three points during the study
* Complete health and lifestyle questionnaires
* Get body composition scans (DEXA) before, during, and after the study

This study may help researchers find new ways to personalize exercise plans based on gut health and improve blood sugar control.

DETAILED DESCRIPTION:
This is a single-arm, interventional study investigating the role of the gut microbiome in mediating the effects of cardiovascular exercise on insulin sensitivity in adult males with overweight or obesity (BMI ≥25). The study also evaluates the effectiveness of sodium butyrate supplementation in enhancing insulin sensitivity among individuals who are otherwise non-responsive to exercise alone.

The study will enroll 25 male participants between the ages of 18 and 40, who are affiliated with Texas Christian University (students, staff, or faculty) and have been sedentary for at least six months. Exclusion criteria include a diagnosis of diabetes or hypertension, recent weight changes, use of antibiotics, probiotics, or weight loss supplements, and any condition contraindicating safe participation in exercise.

Participants will engage in a 12-week supervised cardiovascular exercise program at the TCU Recreation Center. Exercise will progress from 30 to 60 minutes per session, 5 days per week, with intensity increasing from 50% to 80% of estimated maximum heart rate. During weeks 8 through 12, participants will take sodium butyrate (BodyBio; 939 mg sodium/day) in capsule form, dosed at 2 capsules with each meal (6 total/day).

Data collection includes:

* Stool samples (3 total): collected pre-intervention, at week 8 (pre-supplementation), and at week 12 (post-supplementation), to evaluate changes in gut microbial composition and diversity.
* Blood samples (3 total): fasting blood draws at the same three time points to measure glucose and insulin for calculation of HOMA-IR and other insulin sensitivity indices.
* Body composition: assessed at three time points using Dual-Energy X-ray Absorptiometry (DEXA) to determine fat mass, lean mass, and bone mineral density.
* Questionnaires: validated instruments assessing physical activity, dietary intake, sleep, anxiety, depression, and food cravings.

The primary outcomes include changes in insulin sensitivity and gut microbiota composition across the 12-week intervention. Secondary outcomes include body composition changes and the classification of participants as "responders" or "non-responders" to exercise based on insulin sensitivity improvements.

An exploratory objective is to develop predictive models using AI algorithms (e.g., decision trees, random forests, support vector machines, logistic regression) trained on baseline gut microbiota and blood biomarkers to predict individual response to exercise.

This study is internally funded by a TCU Innovation Scholars (IS) Grant (~$20,000), with an in-kind supplement donation valued at $2,000 provided by BodyBio. The study is conducted entirely on the TCU campus and has been approved by the TCU Institutional Review Board (IRB #2025-217). Results from this study aim to advance personalized exercise strategies and contribute to the growing field of precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 to 40 years
* BMI ≥ 25.0 kg/m² (classified as overweight or obese)
* Affiliated with TCU (student, staff, or faculty)
* Sedentary lifestyle, defined as:
* Less than 150 minutes/week of moderate-intensity aerobic activity
* Less than 75 minutes/week of vigorous-intensity activity
* Fewer than 1 strength training session/week over the past 6 months
* Willingness to maintain current diet throughout the study
* Able and willing to understand and complete forms in English
* Able to provide informed consent

Exclusion Criteria:

* Diagnosis of diabetes or currently prescribed insulin
* Hypertension, defined as:
* A diagnosis of high blood pressure
* Currently taking antihypertensive medication
* Blood pressure ≥130/80 mmHg during screening (Visit 1)
* Regular physical activity as defined in inclusion criteria
* Recent significant weight change (≥5% of body weight lost or gained in the past 3 months)
* Use of antibiotics or probiotics in the past 3 months
* Pregnant or planning pregnancy during the study period
* Currently lactating
* Following a restrictive diet (e.g., vegetarian, vegan, keto, carnivore)
* Taking weight loss medications or supplements (e.g., GLP-1 receptor agonists)
* Smoking or excessive alcohol use (>14 drinks/week for men)
* Participation in another research study (clinical trial or intervention study)
* Contraindications to exercise as determined by the Physical Activity Readiness Questionnaire Plus (PARQ+)
* Inability to understand or complete forms in English

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Biological Male Participants
Enrollment: 25 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Change in Insulin Sensitivity (HOMA-IR) | Measured at Baseline (Week 0), Week 8 (pre-supplementation), and Week 12 (post-supplementation)
  Fasting blood glucose and insulin levels will be used to calculate the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR). This outcome will assess the impact of exercise and sodium butyrate supplementation on insulin sensitivity.

SECONDARY OUTCOMES:
Alpha Diversity | Collected at Baseline (Week 0), Week 8, and Week 12
  16S rRNA sequencing of stool samples will be used to evaluate changes in gut microbial alpha diversity in response to exercise and butyrate supplementation.
Lean Mass | Measured at Baseline (Week 0), Week 8, and Week 12
  Dual-Energy X-ray Absorptiometry (DEXA) will assess changes in total lean mass (kg)
Bone mineral density | Measured at Baseline (Week 0), Week 8, and Week 12
  DEXA will be used to measure bone mineral density (g/cm2)
Fat Mass | Measured at Baseline (Week 0), Week 8, and Week 12
  Dexa will be used to measure total fat mass (kg)
Beta diversity | Measured at Baseline (Week 0), Week 8, and Week 12
  16S rRNA sequencing of stool samples will be used to evaluate changes in gut microbial beta diversity in response to exercise and butyrate supplementation.
Taxonomic Classification | Measured at Baseline (Week 0), Week 8, and Week 12
  16S rRNA sequencing of stool samples will be used to evaluate changes in gut microbial taxonomic composition in response to exercise and butyrate supplementation.

OTHER OUTCOMES:
Prediction Accuracy of AI Models for Exercise Response | Modeling conducted post-study using baseline, Week 8, and Week 12 data
  Machine learning algorithms (e.g., random forest, SVM, logistic regression) will be used to predict individual responsiveness to exercise based on baseline gut microbiome and biomarker data. Model performance will be evaluated using classification accuracy, sensitivity, specificity, and AUC.
Anxiety levels | Completed at Baseline (Week 0), Week 8, and Week 12
  Anxiety will be measured through the Beck Anxiety Inventory (BAI). The BAI is a 21-item self-report questionnaire designed to measure the severity of anxiety symptoms, with each item scored on a scale from 0 (not at all) to 3 (severely). Total scores range from 0 to 63, and a higher score indicates more severe anxiety. Specifically, scores of 0-7 reflect minimal anxiety, 8-15 indicate mild anxiety, 16-25 suggest moderate anxiety, and 26-63 signify severe anxiety. Therefore, a higher value on the BAI corresponds to worse anxiety symptoms, providing a clear measure of an individual's anxiety level.
Depression levels | Measured at Baseline (Week 0), Week 8, and Week 12
  Depression will be assessed through the Beck Depression Inventory (BDI). The BDI is a 21-item self-report questionnaire used to assess the severity of depressive symptoms, with each item scored on a scale from 0 (not at all) to 3 (severe). Total scores range from 0 to 63, where a higher score indicates more severe depression. Specifically, scores of 0-13 reflect minimal depression, 14-19 indicate mild depression, 20-28 suggest moderate depression, and 29-63 signify severe depression. Thus, a higher value on the BDI corresponds to worse depressive symptoms, providing a clear measure of an individual's depression level.
Sleep Quality | Measured at Baseline (Week 0), Week 8, and Week 12
  Sleep quality will be measured through the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-item self-report questionnaire designed to assess sleep quality and disturbances over a one-month period. It evaluates seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored from 0 (no difficulty) to 3 (severe difficulty), and the scores are summed to produce a global score ranging from 0 to 21. A higher global score indicates worse sleep quality, with a score of 5 or above typically suggesting poor sleep quality. Thus, a higher value on the PSQI corresponds to greater sleep difficulties, providing a comprehensive measure of an individual's sleep health.
Food reward | Measured at Baseline (Week 0), Week 8, and Week 12
  Food reward will be assessed through the Reward-based Eating Drive scale (RED-13). RED-13 is a 13-item self-report questionnaire designed to assess reward-related eating behaviors, focusing on three key dimensions: lack of control over eating, lack of satiety, and preoccupation with food. Each item is scored to evaluate the intensity of these behaviors, with higher total scores indicating greater reward-driven eating tendencies. The RED-13 is positively associated with body mass index (BMI), food cravings, and self-reported type 2 diabetes diagnosis, making it a valuable tool for identifying individuals with problematic eating patterns. Thus, a higher score on the RED-13 reflects more pronounced reward-based eating behaviors, providing insight into the psychological and physiological drivers of food consumption.
Food consumption | 3 food logs will be applied at Baseline (Week 0), Week 8, and Week 12
  24h food logs will be implemented throughout the study to analyze whether individuals change their diets.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We plan to conduct additional analyses using the samples and data collected in this study beyond the primary aims described in this trial. However, if no further use is identified after the study and initial data analysis are complete, individuals may request information about data sharing by contacting Dr. Elisa Marroquín.

REFERENCES:
- [Background] Noone J, Mucinski JM, DeLany JP, Sparks LM, Goodpaster BH. Understanding the variation in exercise responses to guide personalized physical activity prescriptions. Cell Metab. 2024 Apr 2;36(4):702-724. doi: 10.1016/j.cmet.2023.12.025. Epub 2024 Jan 22. PMID 38262420
- [Background] Cleophas MCP, Ratter JM, Bekkering S, Quintin J, Schraa K, Stroes ES, Netea MG, Joosten LAB. Effects of oral butyrate supplementation on inflammatory potential of circulating peripheral blood mononuclear cells in healthy and obese males. Sci Rep. 2019 Jan 28;9(1):775. doi: 10.1038/s41598-018-37246-7. PMID 30692581
- [Background] Krauze W, Busz N, Pikula W, Maternowska M, Prowans P, Maciejewska-Markiewicz D. Effect of Sodium Butyrate Supplementation on Type 2 Diabetes-Literature Review. Nutrients. 2025 May 22;17(11):1753. doi: 10.3390/nu17111753. PMID 40507022
- [Background] Liu Y, Wang Y, Ni Y, Cheung CKY, Lam KSL, Wang Y, Xia Z, Ye D, Guo J, Tse MA, Panagiotou G, Xu A. Gut Microbiome Fermentation Determines the Efficacy of Exercise for Diabetes Prevention. Cell Metab. 2020 Jan 7;31(1):77-91.e5. doi: 10.1016/j.cmet.2019.11.001. Epub 2019 Nov 27. PMID 31786155
- [Background] Boule NG, Weisnagel SJ, Lakka TA, Tremblay A, Bergman RN, Rankinen T, Leon AS, Skinner JS, Wilmore JH, Rao DC, Bouchard C; HERITAGE Family Study. Effects of exercise training on glucose homeostasis: the HERITAGE Family Study. Diabetes Care. 2005 Jan;28(1):108-14. doi: 10.2337/diacare.28.1.108. PMID 15616242
- [Background] Bohm A, Weigert C, Staiger H, Haring HU. Exercise and diabetes: relevance and causes for response variability. Endocrine. 2016 Mar;51(3):390-401. doi: 10.1007/s12020-015-0792-6. Epub 2015 Dec 7. PMID 26643313